CLINICAL TRIAL: NCT01586377
Title: Near-infrared Spectroscopic Measurement of Tissue Oxygen Saturation and the Vascular Occlusion Test in Complex Regional Pain Syndrome
Brief Title: Near-infrared Spectroscopic Measurement in Complex Regional Pain Syndrome
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Geoff Bellingham, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-11-382; 18119 (Other: Research Ethics Board number)
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Reflex Sympathetic Dystrophy
Keywords: Complex regional pain syndrome; Near Infrared Spectroscopy; Vascular Occlusion Test
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CRPS Type 1: Patients with CRPS 1 affecting a single upper limb
- Healthy volunteers: Volunteers without the diagnosis of CRPS Type 1

SUMMARY:
Recent clinical investigations have suggested that the cause of abnormal pain in complex regional pain syndrome could be ischemia and inflammation, due to poor blood flow to deep tissues from microvascular pathology. This study aims to determine if a new technology called near infrared spectroscopy can measure this microvascular dysfunction. The study hypothesizes that significant differences can be measured in the microcirculation of patients with CRPS-I using near infrared spectroscopy and the vascular occlusion test.

DETAILED DESCRIPTION:
The pathophysiology of CRPS-1 is unknown yet a considerable number of studies suggest that the fundamental cause of abnormal pain is due to microvascular pathology of deep tissues.

Reduced blood flow to deep tissues such as muscle, nerve, and bone can lead to a combination of inflammatory and neuropathic pain processes (Coderre TJ et al. 2010). Evidence to support this model of microcirculatory dysfunction includes observations that skin capillary oxygenation is decreased and skin lactate is increased in affected limbs of patients (total of 11 patients in lactate study) (Birklein F et al. 2000, Manahan AP et al. 2007). It has also been reported that patients with CRPS-I have abnormal vasodilatory responses after sympathetically-mediated vasoconstriction (Dayan L et al. 2008) and decreased concentrations of nitric oxide in the affected limb (Groeneweg JG et al. 2006).

Near-infrared spectroscopy (NIRS) is a non-invasive method of measuring tissue oxygenation using the differential absorption properties of oxygenated and deoxygenated hemoglobin in biological tissue (Creteur J 2008). Near-infrared light is only transmitted through small vessels with diameter less than 1 mm (arterioles, venules and capillaries). Since NIRS is limited to monitoring only small vessels, it can be used to assess oxygen balance in the microcirculation of skeletal muscle (Creteur J 2008).

Premises Premise 1: Complex regional pain syndrome is associated with microcirculatory dysfunction

After an injury to a patient's limb, it is hypothesized that the pressure exerted by that swelling within a relatively confined anatomical space can occlude the capillaries of adjacent tissues and cause a compartment syndrome-like injury. Coderre et al. (2010) have theorized that the resulting microcirculatory dysfunction causes a persistent inflammatory state which is then responsible for pain generation.

In an animal model of ischemia-reperfusion injury used to study CRPS-1, microscopy of muscle and nerve tissue demonstrates microvascular evidence of a slow-flow/no-reflow phenomenon (Coderre TJ et al. 2010). Existence of a slow-flow/no-reflow state causes persistent inflammation in deep tissue. Animals subsequently develop hyperemia and edema, followed by mechano-hyperalgesia, allodynia, and cold-allodynia lasting for at least 1 month (Coderre et al. 2010). This clinical picture is similar to the clinical signs of those patients afflicted with CRPS-1.

Premise 2: Vascular occlusion testing measures microcirculatory dysfunction NIRS measurement of peripheral tissue oxygen saturation (StO2), combined with a reproducible ischemia-reperfusion challenge to induce reactive hyperemia (vascular occlusion testing - VOT), has been described as a valid and reliable method for assessing microcirculatory dysfunction (De Backer et al. 2010). This involves a short period of forearm ischemia by inflating a blood pressure cuff on the upper arm. The blood pressure cuff is then released after approximately 3 minutes and this followed by reperfusion of the forearm. This stimulates the release of endogenous nitric oxide (NO) from the microvascular endothelium (Harel et al 2008). Measurement of this hyperemic response using NIRS has been demonstrated to be a feasible non-invasive method of quantifying microcirculatory function. This technique shares strong correlation with the gold-standard method of strain gauge plethysmography (Harel et al. 2008).

ELIGIBILITY:
Inclusion Criteria:

* Complex regional pain syndrome type 1 (CRPS-I) of one upper extremity.
* Healthy volunteers.
* Diagnosis of CRPS-I established for greater than 12 weeks.

Exclusion Criteria:

* Pregnancy
* Lack of informed consent
* History of peripheral vascular disease requiring angioplasty or bypass surgery
* History of systemic vasculitis
* Current use of vasoactive medications
* Diabetes Type I and II
* Presently smoking

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CRPS Type 1 will be selected from a tertiary care chronic pain clinic. Healthy volunteers will be selected from a community sample
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Baseline tissue oxygen saturation | Day 1

SECONDARY OUTCOMES:
Occlusion slope during vascular occlusion test | Day 1
Reperfusion slope during vascular occlusion test | Day 1
Delta StO2 | Day 1
  Defined as the difference between the maximal tissue oxygenation value after reperfusion and the baseline measurement
Post-obstructive hyperemic response | Day 1
Thenar muscle oxygen consumption | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Geoff A Bellingham, MD FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- Pain Clinic, St. Joseph's Health Care London Hospitals, London, Ontario, Canada

REFERENCES:
- [Background] Birklein F, Weber M, Neundorfer B. Increased skin lactate in complex regional pain syndrome: evidence for tissue hypoxia? Neurology. 2000 Oct 24;55(8):1213-5. doi: 10.1212/wnl.55.8.1213. PMID 11071503
- [Background] Creteur J. Muscle StO2 in critically ill patients. Curr Opin Crit Care. 2008 Jun;14(3):361-6. doi: 10.1097/MCC.0b013e3282fad4e1. PMID 18467900
- [Background] Coderre TJ, Bennett GJ. A hypothesis for the cause of complex regional pain syndrome-type I (reflex sympathetic dystrophy): pain due to deep-tissue microvascular pathology. Pain Med. 2010 Aug;11(8):1224-38. doi: 10.1111/j.1526-4637.2010.00911.x. PMID 20704671
- [Background] Dayan L, Salman S, Norman D, Vatine JJ, Calif E, Jacob G. Exaggerated vasoconstriction in complex regional pain syndrome-1 is associated with impaired resistance artery endothelial function and local vascular reflexes. J Rheumatol. 2008 Jul;35(7):1339-45. Epub 2008 May 1. PMID 18464300
- [Background] De Backer D, Ospina-Tascon G, Salgado D, Favory R, Creteur J, Vincent JL. Monitoring the microcirculation in the critically ill patient: current methods and future approaches. Intensive Care Med. 2010 Nov;36(11):1813-25. doi: 10.1007/s00134-010-2005-3. Epub 2010 Aug 6. PMID 20689916
- [Background] Doerschug KC, Delsing AS, Schmidt GA, Haynes WG. Impairments in microvascular reactivity are related to organ failure in human sepsis. Am J Physiol Heart Circ Physiol. 2007 Aug;293(2):H1065-71. doi: 10.1152/ajpheart.01237.2006. Epub 2007 May 4. PMID 17483235
- [Background] Groeneweg JG, Huygen FJ, Heijmans-Antonissen C, Niehof S, Zijlstra FJ. Increased endothelin-1 and diminished nitric oxide levels in blister fluids of patients with intermediate cold type complex regional pain syndrome type 1. BMC Musculoskelet Disord. 2006 Nov 30;7:91. doi: 10.1186/1471-2474-7-91. PMID 17137491
- [Background] Harel F, Denault A, Ngo Q, Dupuis J, Khairy P. Near-infrared spectroscopy to monitor peripheral blood flow perfusion. J Clin Monit Comput. 2008 Feb;22(1):37-43. doi: 10.1007/s10877-007-9105-9. Epub 2007 Nov 27. PMID 18040873
- [Background] Skarda DE, Mulier KE, Myers DE, Taylor JH, Beilman GJ. Dynamic near-infrared spectroscopy measurements in patients with severe sepsis. Shock. 2007 Apr;27(4):348-53. doi: 10.1097/01.shk.0000239779.25775.e4. PMID 17414414
- [Derived] Bellingham GA, Smith RS, Morley-Forster P, Murkin JM. Use of near infrared spectroscopy to detect impaired tissue oxygen saturation in patients with complex regional pain syndrome type 1. Can J Anaesth. 2014 Jun;61(6):563-70. doi: 10.1007/s12630-014-0140-y. Epub 2014 Mar 26. PMID 24668314